CLINICAL TRIAL: NCT06736054
Title: A Phase I Trial of 61Cu-NODAGA-PSMA for Patients with Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 189-21-CA
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Prostate Adenocarcinoma
Keywords: PSMA; PET/CT; Phase 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prostate Adenocarcinoma with PSMA-Positive Disease on a PSMA Targeted PET/CT (Experimental): TEST PRODUCT, DOSE, AND ROUTE OF ADMINISTRATION: Subjects will undergo imaging with 100-300 MBq (2.7-8.1 mCi) of 61Cu-NODAGA-PSMA intravenously (IV), followed by PET/CT imaging 60 (+/- 10) minutes post radiotracer administration.
  Interventions: Drug: Copper 61-PSMA PET/CT

INTERVENTIONS:
Drug: Copper 61-PSMA PET/CT — TEST PRODUCT, DOSE, AND ROUTE OF ADMINISTRATION: Subjects will undergo imaging with 100-300 MBq (2.7-8.1 mCi) of 61Cu-NODAGA-PSMA intravenously (IV), followed by PET/CT imaging 60 (+/- 10) minutes post radiotracer administration.

SUMMARY:
Molecular Imaging (MI) uses tracers which emit radiation to provide clinically valuable imaging for patient with cancer. Most current MI agents utilize Fluorine 18 or Gallium 68 as the positron emitter for PET imaging. However, these isotopes have short half-lives which limit the geographic distribution range of tracers made with these isotopes. Copper 61 (61Cu) has a 3.3 hour half-life, which would allow for far greater distribution range following radiotracer production.

This phase I trial will test the safety and effectiveness of a novel MI radiotracer that uses 61Cu as its positron emitting isotope and targets Prostate Specific Membrane Antigen (PSMA) for imaging prostate cancer. A successful trial will provide the ability to advance this novel 61Cu-NODAGA-PSMA radioisotope into phase II trials, as well as open a new paradigm into the production of MI radioisotopes with 61Cu.

DETAILED DESCRIPTION:
This is a phase 1, non-randomized study. Subjects will undergo imaging with 100-300 MBq (2.7-8.1 mCi) of 61Cu-NODAGA-PSMA intravenously (IV), followed by PET/CT imaging 60 (+/- 10) minutes post radiotracer administration. This is a diagnostic imaging study. As the imaging agent will not have a treatment effect, efficacy evaluations that are standard in treatment protocols will not be performed. We expect to enroll 6-10 patients in the proposed study. The sample size is exploratory.

For the primary objective of safety, side effects will be monitored the day of and the day following radiotracer administration. As the PET radiotracer used in this trial is given at a low, imaging dose, serious adverse events are not expected. If a single serious adverse event is identified, then the protocol will be held until reviewed by the IRB.

For the secondary objective of dosimetry, dosimetry will be calculated from PET/CT images and radioactive counts in blood samples by an experience medical physicist.

For the secondary objective of effectiveness, the number of suspected PSMA-positive malignant lesions will be calculated in both the standard-of-care 18F-Piflufolastat PET/CT and the experimental 61Cu- PSMA PET/CT. Positive lesions will be considered to be the foci greater than local background that are not physiologic/benign by location. The percentage of patients with any suspected PSMApositive malignant lesions will be determined for each radiotracer.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven prostate adenocarcinoma
2. Age ≥ 18 years
3. ECOG 0 or 1
4. At least one site of PSMA-positive disease on a PSMA-targeted PET/CT performed within 30 days of trial recruitment
5. Creatinine of ≤1.4 or Creatinine Clearance or ≥ 60 mL/minute.

Exclusion Criteria:

1. Known allergy/hypersensitivity to PSMA-targeted imaging agents
2. Other active malignancy, other than the known prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Imaging Agent-Emergent Adverse Events [Safety and Tolerability] | Up to 24 hours after administration of radiotracer
  For the primary objective of safety, side effects will be monitored the day of and the day following radiotracer administration.

SECONDARY OUTCOMES:
Dosimetry | Up to 24 hours after administration of radiotracer
  For the secondary objective of dosimetry, dosimetry will be calculated from PET/CT images and radioactive counts in blood samples by an experience medical physicist.
Number of suspected PSMA-positive malignant lesions | Up to 24 hours after administration of radiotracer
  For the secondary objective of effectiveness, the number of suspected PSMA-positive malignant lesions will be calculated in both the standard-of-care 18F-Piflufolastat PET/CT and the experimental 61Cu-PSMA PET/CT. Positive lesions will be considered to be the foci greater than local background that are not physiologic/benign by location. The percentage of patients with any suspected PSMA-positive malignant lesions will be determined for each radiotracer.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Basaco Bernabeu T, Mansi R, Del Pozzo L, Zanger S, Gaonkar RH, McDougall L, De Rose F, Jaafar-Thiel L, Herz M, Eiber M, Ulaner GA, Weber WA, Fani M. 61Cu-PSMA-Targeted PET for Prostate Cancer: From Radiotracer Development to First-in-Human Imaging. J Nucl Med. 2024 Sep 3;65(9):1427-1434. doi: 10.2967/jnumed.123.267126. PMID 39025646